CLINICAL TRIAL: NCT05501769
Title: A Phase 1b Trial of ARV-471 in Combination With Everolimus in Patients With ER+, HER2- Advanced or Metastatic Breast Cancer
Brief Title: ARV-471 in Combination With Everolimus for the Treatment of Advanced or Metastatic ER+, HER2- Breast Cancer
Acronym: TACTIVE-E
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arvinas Estrogen Receptor, Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Arvinas Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARV-471-mBC-102; C4891020 (Other: Pfizer)
Record Dates: First submitted 2022-08-09; First posted 2022-08-15 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Advanced breast cancer; Metastatic breast cancer; MBC; Endocrine therapy; Estrogen receptor; ER+; human epidermal growth factor receptor 2; HER2-; ARV-471; Everolimus; PROTAC; Vepdegestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ARV-471 and Everolimus (Experimental): ARV-471 oral tablets in combination with everolimus administered daily in 28 day cycles
  Interventions: Drug: ARV-471 in combination with Everolimus

INTERVENTIONS:
Drug: ARV-471 in combination with Everolimus — ARV-471 oral tablets in combination with everolimus administered daily in 28 day cycles

SUMMARY:
A phase 1b study to assess the combination of ARV-471 and everolimus in participants with advanced or metastatic ER+/HER2- breast cancer.

DETAILED DESCRIPTION:
This is a Phase 1b study to assess the safety and tolerability of ARV-471 in combination with everolimus in participants with estrogen receptor positive/human epidermal growth factor receptor 2 negative (ER+/HER2-) advanced or metastatic breast cancer, who have received a prior CDK4/6 inhibitor and endocrine therapy in the advanced/metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ER+ and HER2-advanced breast cancer (metastatic, recurrent, or unresectable)
* Women must be postmenopausal, or pre-/peri-menopausal women must be on ovarian suppression
* Measurable disease or non-measurable (evaluable) disease per RECIST v1.1
* Received a minimum of 1 and up to 3 lines of anti-cancer therapy in the advanced/metastatic setting: must have received and progressed on (or were intolerant to) a CDK 4/6 inhibitor, either alone or in combination; must have received at least one endocrine therapy, either alone or in combination; may have received up to one line of chemotherapy
* Must be willing to use dexamethasone mouthwash for the prevention of everolimus-induced stomatitis
* ECOG performance status of 0 or 1

Exclusion Criteria:

* Untreated brain metastases or brain metastases requiring steroids above physiologic replacement doses
* Prior treatment with ARV-471
* Prior treatment targeting mTOR (e.g. everolimus)
* Prior anticancer or investigational drug treatment within 28 days (fulvestrant) or 14 days (tamoxifen or aromatase inhibitor, or CDK 4/6 inhibitor) before the first dose of study drug
* Prior anticancer or investigational anticancer drug therapy within 28 days or 5 half-lives (whichever is shorter) before the first dose of study drug, except as mentioned above
* Any of the following in the previous 12 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, symptomatic pulmonary embolism, or other clinically significant episode of thromboembolism
* Any of the following in the previous 6 months: congenital long QT syndrome, Torsade de Pointes, sustained ventricular tachyarrhythmia and ventricular fibrillation, left anterior hemiblock, ongoing cardiac arrythmias/dysrhythmias, atrial fibrillation
* Hypertension that cannot be controlled by medication (>150/90 mmHg despite optimal medical therapy)
* Active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus, hepatitis C virus, known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness
* Known history of drug-induced pneumonitis or other significant symptomatic deterioration of lung function
* Live vaccines within 14 days before the first dose of study drug
* Major surgery (as defined by the Investigator) within 4 weeks of first dose of study drug
* Radiation therapy within 4 weeks of first dose of study drug or prior irradiation to more than 25% of the bone marrow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-09-08 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities of ARV-471 in combination with everolimus | 35 Days
  Dose limiting toxicities in the first 35 days of the study combination treatment characterized by type, frequency, severity (as graded by NCI CTCAE v5.0), timing, seriousness, and relationship to study drug
Recommended Phase 2 Dose (RP2D) for ARV-471 in combination with everolimus | 35 Days
Number of participants with adverse events as a measure of safety and tolerability of ARV-471 in combination with everolimus | 28 calendar days after participant discontinues study treatment
  Adverse events as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study drug combination
Incidence of laboratory abnormalities as a measure of safety and tolerability of ARV-471 in combination with everolimus | 28 calendar days after participant discontinues study treatment
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v5.0), and timing

SECONDARY OUTCOMES:
Overall response rate (ORR) in participants | Up to approximately 1 year
Clinical benefit rate (CBR) in participants. | Up to approximately 1 year
  Clinical benefit response rate based on the summation of CRs, PRs and stable disease of 24 weeks duration or longer.
Duration of response (DOR) in participants | Up to approximately 1 year
Maximum plasma concentrations (Cmax) of ARV-471 and everolimus | At predefined intervals throughout the treatment period, up to approximately 4 weeks after last dose of investigational products
Time to maximum plasma concentrations (Tmax) of ARV-471 and everolimus | At predefined intervals throughout the treatment period, up to approximately 4 weeks after last dose of investigational products
Area under the concentration-time curve over 24 hours at steady state (AUC(0-24)) of ARV-471 and everolimus | At predefined intervals throughout the treatment period, up to approximately 4 weeks after last dose of investigational products

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, Santa Monica, California
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Lake Mary, Florida
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, Nashville, Tennessee
- Spain (3):
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Valencia

IPD SHARING:
Plan to Share IPD: No